CLINICAL TRIAL: NCT07039656
Title: Toripalimab Combined With Chemotherapy as Postoperative Adjuvant Therapy for Non-Small Cell Lung Cancer With or Without Prior Neoadjuvant Therapy: A Two-Cohort, Multicenter Phase II Trial
Brief Title: Toripalimab Combined With Chemotherapy as Adjuvant Therapy for Non-small Cell Lung Cancer With or Without Prior Neoadjuvant Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wen-zhao ZHONG (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor-Investigator, Wen-zhao ZHONG, Head of Thoracic Surgery, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-1057-03
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-06

CONDITIONS: Stage IB-IIIB NSCLC; Stage IIB-III NSCLC
Keywords: Toripalimab; MRD; Adjuvant therapy
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage IB-IIIB participants following completely resection without neoadjuvant therapy (Experimental)
  Interventions: Drug: Toripalimab; Drug: Cisplatin-based chemotherapy
- Stage IIB-III participants with non-MPR or MPR but lymph node positivity after neoadjuvant therapy (Experimental)
  Interventions: Drug: Toripalimab; Drug: Cisplatin-based chemotherapy

INTERVENTIONS:
Drug: Toripalimab — Participants will receive Toripalimab (240 mg IV) Q3W for 17 cycles (cycle length=21 days).
Drug: Cisplatin-based chemotherapy — Cisplatin[75 mg/m^2 IV Q3W]/carboplatin[AUC 5 IV Q3W]+paclitaxel[260 mg/m^2 IV Q3W] or cisplatin[75 mg/m^2 IV Q3W)]/carboplatin[AUC 5 IV Q3W]+ pemetrexed[500 mg/m2 IV Q3W],dependent on tumor histology. Participants will receive Chemotherapy for 3-4 cycles

SUMMARY:
This is a two-cohort, multicenter, Phase II study to evaluate the efficacy and safety of 3-4 cycles of toripalimab (JS001) plus chemotherapy followed by toripalimab maintenance treatment up to one year in participants with completely resected non-small cell lung cancer (NSCLC) stratified by prior neoadjuvant treatment status, as measured by disease-free survival (DFS) and overall survival (OS).

Researchers will compare outcomes between two cohorts:

1. Cohort 1: Stage IB-IIIB participants following completely resection without neoadjuvant therapy;
2. Cohort 2: Stage IIB-III participants with non-MPR or MPR but lymph node positivity after neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Patient with age ≥ 18 and ≤75 years old, gender is not limited.
3. Cohort 1: Histological diagnosis of Stage IB -IIIB NSCLC without anti-cancer treatment; Cohort 2: Histological diagnosis of Stage IIB-III NSCLC with non-MPR or MPR but lymph node positivity after neoadjuvant chemoimmunotherapy; (per American Joint Committee on Cancer staging system (AJCC) staging system, 8th edition)
4. Participants must have had complete resection of NSCLC 60 days
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
6. Adequate organ function performed within 10 days of treatment initiation
7. Male or female patients of childbearing potential will voluntarily use an effective method of contraception, e.g., double-barrier contraception, condoms, oral or injectable contraceptives, IUDs, etc., during the study period and for the last 6 months of study drug use. All female patients will be considered of childbearing potential unless the female patient is naturally menopausal, artificially menopausal or sterilised (e.g. hysterectomy, bilateral adnexectomy or radiation ovarian irradiation).

Exclusion Criteria:

1. Pathological histology confirmed the diagnosis of small cell lung cancer pathological type;
2. Treatment with prior systemic chemotherapy at any time
3. Confirmed EGFR or ALK mutations
4. Patient has a history of active autoimmune disease or autoimmune disease that may recur
5. Active hepatitis B and C patients will need to be on relevant antiviral therapy, have HBV-DNA <2000 IU/ml (<104 copies/ml) and have received anti-HBV therapy for at least 14 days prior to study participation, and continue therapy for the duration of the treatment period; HCV RNA-positive patients must be on antiviral therapy and have a liver function that is within the elevated CTCAE grade 1;
6. Known allergy to chemotherapy drugs including cisplatin, paclitaxel, albumin-paclitaxel and pemetrexed;
7. History of allergy to monoclonal antibody drugs
8. Patients with previous allogeneic stem cell or parenchymal organ transplantation
9. Having a mental illness or any other condition that renders treatment non-compliant
10. Patients unable or unwilling to sign the informed consent form
11. The investigator considered that the patient's condition may affect compliance with the protocol or make participation in this study unsuitable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year Disease-Free Survival | 24 months
  DFS was defined as the time from the start of the treatment to either the date of disease recurrence or death (whatever the cause) as assessed by the investigator. Recurrence of disease was defined as local regional recurrence, a distant (metastatic) recurrence, or a second primary cancer. Occurrence of a second extra-pulmonary malignancy was considered to be an event.

SECONDARY OUTCOMES:
Overall Survival | 60 months
  OS was defined as the time from the start of treatment to the date of death.
Adverse events | 24 months
  Incidence of AE/SAE which has been confirmed correlation with treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Treatment and survival data for participants will be presented in the corresponding manuscript.